CLINICAL TRIAL: NCT06578312
Title: A Study on Establishing a "Critical State" Early Warning Score After Congenital Heart Disease Surgery and an Integrated Treatment Model of a Multidisciplinary Rapid Response Team
Brief Title: "Critical State" Early Warning Score After CHD Surgery and Rapid Response Team
Status: Completed | Type: Observational
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Xu Wang, Chief Physician, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 2022-GSP-GG-32
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Congenital Heart Disease
Keywords: congenital heart disease; Early warning system; machine learning; retrospective study
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
By establishing a warning scoring tool for the early "critical state" after congenital heart disease surgery, the multidisciplinary rapid response team is proactively activated, forming an integrated treatment model of early warning-team decision-making-organ assistance.

DETAILED DESCRIPTION:
All children aged 0-14 years admitted to the PICU from 2021-2022 were enrolled continuously, and their baseline data such as gender, age, RACHS-1 score, cardiopulmonary bypass time, aortic clamping time, whether there was chromosomal lesions, whether there was preoperative endotracheal intubation/heart failure, changes in oxygenation index, lactate, and vasoactive drug scores were obtained. All variables that may lead to composite malignant events including death in the early postoperative period were included, including death, pulmonary hypertension crisis, malignant arrhythmias (supraventricular tachycardia, ventricular tachycardia, ventricular fibrillation, high-degree atrioventricular block) requiring antiarrhythmic drugs or pacemaker treatment, cardiopulmonary resuscitation, ECPR, emergency sternal expansion, severe AKI, severe ARDS, neurological complications (cerebral hemorrhage, cerebral infarction), gastrointestinal complications (gastrointestinal bleeding, intestinal obstruction, intestinal necrosis).The variables were included in the machine learning analysis to establish the model.

ELIGIBILITY:
Inclusion Criteria:

* pediatrics admitted to ICU

Exclusion Criteria:

* surgery without cardiopulmonary bypass
* neonatal
* using extra-corporeal circulation during surgery
* Delayed chest closing during surgery

Ages: 28 Days to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: We included pediatrics with congenital heart disease who undergone surgery in our center.They should under 14 years old.
Sampling Method: Non-Probability Sample
Enrollment: 4115 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
event occurrence-an inclusion of composite clinical diagnose | Within 48 hours after surgery
  critical status included clinical diagnose：arrhythmia（ventricular tachycardia、ventricular fibrillation、refractory supraventricular tachycardia
  ）,prognosis（death or live）,bedside thoracotomy,CPR,ECMO,extracorporeal circulation establishment,renal replacement therapy,peritoneal dialysis, hemofiltration. If one of the above diagnosis and treatment used in patients, they would be divided to case group.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Wang, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
It included some private information.